CLINICAL TRIAL: NCT03619122
Title: Impact of Second Forward View Examination of Proximal Colon on Adenoma Detection Rate: A Randomized Clinical Trial
Brief Title: Second Forward View Examination of Proximal Colon on Adenoma Detection Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2018-R014
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Colon Adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second Examination (Experimental): Eligible patients who consent to participate undergo planned colonoscopy by endoscopists performing procedures that day per normal standard of care. The colonoscope is passed to the cecum and then withdrawn to the hepatic flexure with washing and aspirating of colonic contents as needed to optimize visualization of colonic mucosa. Then, the colonoscope is inserted to the cecum and withdrawn to the hepatic flexure again for second examination.
  Interventions: Procedure: Second Examination
- Traditional Examinaiton (No Intervention): Eligible patients who consent to participate undergo planned colonoscopy by endoscopists performing procedures that day per normal standard of care. The colonoscope is passed to the cecum and then withdrawn to the hepatic flexure with washing and aspirating of colonic contents as needed to optimize visualization of colonic mucosa. Then, the colonoscope is withdrawn to the anus directly.

INTERVENTIONS:
Procedure: Second Examination — The colonoscopy is passed to the cecum and then withdrawn to hepatic flexure. Then, the scopy is inserted to the cecum and withdrawn to hepatic flexure again for second foreard view examination.
  Arms: Second Examination

SUMMARY:
This clinical trial is being conducted to assess whether second forward view examination of proximal colon could increase adenoma detection rate of right colon.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing colonoscopy for screening in our hospital

Exclusion Criteria:

* previous history of resection of colon;
* familial polyposis syndrome
* inflammatory bowel disease
* active antiplatelet or anticoagulant therapy prevent polypectomy;
* pregnancy or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
per-patient detection rate of adenoma of proximal colon | 1 day
  the number of patients with at least one adenoma identified divided by total number of patients completing colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Shan K, Lu H, Zhang Z, Xie J, Xu L, Wang W, Hu C, Xu L. Impact of second forward-view examination on adenoma detection rate during unsedated colonoscopy: a randomized controlled trial. BMC Gastroenterol. 2021 May 10;21(1):213. doi: 10.1186/s12876-021-01783-9. PMID 33971824